CLINICAL TRIAL: NCT03085511
Title: Does Higher Protein Quality Reduce Energy Intake When Following a Weight Loss Diet Plan? -- Nonpilot, Powered Crossover
Brief Title: High Quality Protein for Assisting With Weight Loss
Acronym: Egg_breakfast
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Collaborators: American Egg Board (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TTU IRB2016-1137
Record Dates: First submitted 2017-03-15; First posted 2017-03-21 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Obesity
Keywords: Egg breakfast; Weight loss; Satiety; Insulin; Glucagon-Like Peptide 1; PYY (3-36) peptide; Ghrelin; Glucose; Protein quality
MeSH Terms: conditions — Obesity; Weight Loss; Insulin Resistance | interventions — Diet, Reducing

STUDY DESIGN:
Intervention Model Description: Within subjects comparison will be performed. Subjects will be assigned to either group A (EB first then CB) or group B (CB first then EB) for a week and then reverse to the opposite breakfast the next week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Egg Breakfast (EB) (Experimental): The EB will receive the following breakfast:
  2 scrambled eggs, 120 mL skim milk, 2 slices of Mrs. Bairds® Extra Thin White Bread, 5 g of butter, and 18 g of Smuckers® Strawberry Jam.
  Interventions: Behavioral: Egg breakfast (EB); Behavioral: Weight Loss Counseling; Behavioral: Weight Loss Diet
- Cereal Breakfast (CB) (Active Comparator): The CB will receive the following breakfast:
  1.5 cups of Special K® Ready-to-Eat Original Cereal, 200 ml Silk® Original Soymilk, 1 slice of Nature's Own® Double Fiber Wheat Bread, 13 g of butter, and 10 g of Smuckers® Sugar-Free Strawberry Jam.
  Interventions: Behavioral: Weight Loss Counseling; Behavioral: Weight Loss Diet; Behavioral: Cereal Breakfast (CB)

INTERVENTIONS:
Behavioral: Egg breakfast (EB) — Breakfast is considered as high quality protein diet, but has similar weight, energy, and macronutrients as the active comparator. The details are as follows: weight 291 g,energy 400 kcal, energy density 1.37 kcal/g, carbohydrate 42.9%, fat 35.6%, protein 19.8%, protein digestibility corrected amino acid score (PDCAAS) 100, leucine 1.77 g, glycemic load 24, fiber 1.0 g.
  Arms: Egg Breakfast (EB)
Behavioral: Weight Loss Counseling — Weight loss counseling will be administered by a Registered Dietitian and will utilize information and materials derived from the Evidence Analysis Library (EAL) of the Academy of Nutrition and Dietetics (AND). Topics will include portion control, macronutrient distribution, snacking, eating out, cooking and grocery shopping, as well as behavioral strategies including self-monitoring, motivational interviewing, goal setting, and problem solving.
Behavioral: Weight Loss Diet — Participants will have a 1200-1500kcals diet based on each individual's body weight during the study.
Behavioral: Cereal Breakfast (CB) — Breakfast is considered as low quality protein diet, but has similar weight, energy, and macronutrients as that in experimental group. The details are as follows: weight 293 g, energy 398 kcal, energy density 1.36 kcal/g, carbohydrate 44.8%, fat 35.4%, protein 19.8%, protein digestibility corrected amino acid score (PDCAAS) 42, leucine 0.48 g, glycemic load 30.8, fiber 4.4 g.
  Arms: Cereal Breakfast (CB)

SUMMARY:
The purpose of this study is to determine if, in presence of a reduced calorie diet, a breakfast containing high quality protein source (eggs) would be more effective in reducing hunger and increasing feeling of fullness compared to a breakfast containing a lower quality of protein, but equal energy density. A previous pilot study with the same endpoints yielded borderline significant results; this study has been powered based on that pilot to interrogate our hypotheses.

DETAILED DESCRIPTION:
This will be a crossover study with 2 experiments. Subjects will follow a reduced energy weight loss diet of 1,200-1,500 kcal adjusted to each individual's body weight for totally 2 weeks in each experiment. They will come to the clinic from day 1 to day 7 and consume egg breakfast (EB) for 5 days under our supervision. Then on weekends during this period they will continue this breakfast at home based on our advice. The next week they will have cereal breakfast (CB) and the process is similar to that in the first week.

The 1st experiment will test the satiety from egg breakfast (EB) and following energy intake in both lunch and dinner, compared with CB (cereal breakfast). Lunch and dinner will be offered on 2 test days during each week. Anthropometric and body composition measurements, blood pressure, blood draw, satiety questionnaire, as well as energy intake will also be collected in the 2 test days and compared between 2 breakfast groups.

The 2nd one is to test whether EB will help in resisting the intake of foods considered tempting, but detrimental to weight loss efforts, compared with CB. The process is similar to experiment 1 except no blood draw, no dinner offered. Instead, a tempting food after lunch will be offered.

ELIGIBILITY:
Inclusion Criteria:

* Overweight and class I-II obese (BMI 25.0-39.9)
* Sedentary (<3 hours/week of moderate intensity physical activity)
* Otherwise healthy

Exclusion Criteria:

* ≥5% body weight loss or gain in the three months preceding the study
* Post-menopausal (has not had period for 12 months)
* Plans to begin an exercise program or change current exercise routines between initiation of study and final study
* Anyone following a medical diet prescription
* Anyone with a chronic disease including type II diabetes, hypothyroidism, hypoparathyroidism, cardiovascular disease, cancer of any type
* Health conditions and chronic illness that contraindicate behavioral weight loss treatment using a low calorie diet: Unstable cardiac condition; Polycystic ovary syndrome; Prader-Willi syndrome; Major systemic illness; History of recreational drug abuse or eating disorder (Binge Eating Disorder); Familial hyperlipidemia; Major endocrine diseases (Cushing's syndrome, Grave's disease, Hashimoto's thyroiditis); Gastrointestinal disorder
* Anyone who is currently pregnant, or lactating
* Medications that may influence or inhibit appetite, sensory functioning, or hormone signaling
* Plans to begin taking any supplements that may influence weight loss
* Report of medical condition or surgical intervention that affects swallowing or chewing ability
* Anyone with a pacemaker or other internal medical device
* Any practicing vegans or vegetarians
* Any practicing gluten-free diet
* Allergy, aversion, or dislike to any of the foods offered for meals

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-08-20 (Actual); Primary Completion 2019-05-17 (Actual); Study Completion 2019-05-17 (Actual)

PRIMARY OUTCOMES:
Change of subjective satiety | Change in scores (arbitrary units AUC) from 30 minutes before breakfast consumption to 240 minutes after the consumption on day 7 and day 14
  This will be measured by questionnaire (VAS) and compared the changes between 2 test days (day 7 and day 14) in experiment 1&2
Change of objective satiety | Change in concentration (AUC) from 30 minutes before breakfast consumption to 180 minutes after the consumption on day 7 and day 14
  It is measured by GLP-1. This will be tested in experiment 1 and changes will be compared between 2 test days.
Change of objective satiety | Change in concentration (AUC) from 30 minutes before breakfast consumption to 180 minutes after the consumption on day 7 and day 14.
  It is measured by PYY 3-36. This will be tested in experiment 1 and changes will be compared between 2 test days.
Change of objective satiety | Change in concentration (AUC) from 30 minutes before breakfast consumption to 180 minutes after the consumption on day 7 and day 14.
  It is measured by ghrelin. This will be tested in experiment 1 and changes will be compared between 2 test days.
Other change of hormone level | Change in concentration (AUC) from 30 minutes before breakfast consumption to 180 minutes after the consumption on day 7 and day 14.
  It is measured by serum glucose. This will be tested in experiment 1 and changes will be compared between 2 test days.
Other change of hormone level | Change in concentration (AUC) from 30 minutes before breakfast consumption to 180 minutes after the consumption on day 7 and day 14.
  It is measured insulin levels. This will be tested in experiment 1 and changes will be compared between 2 test days.
Energy intake (kcal) during ad libitum lunch | Test day 7 and day 14
  Energy intake will be compared between 2 test days in experiment 1
Energy intake (kcal) during ad libitum dinner | Test day 7 and day 14
  Energy intake will be compared between 2 test days in experiment 1
Energy intake (kcal) during ad libitum lunch | Test day 7 and day 14
  Chocolate brownies will be added to the test lunch. Energy intake will be compared between 2 test days in experiment 2

SECONDARY OUTCOMES:
Change in body weight (kg) | Day 0, day 7 and day 14
  Body weight change from baseline to day 7, and change from day 7 to day 14 will be compared
Change in waist and hip circumference (cm) | Day 0, day 7 and day 14
  Waist and hip circumference change from baseline to day 7, and change from day 7 to day 14 will be compared
Change in blood pressure (mm Hg) | Day 0, day 7 and day 14
  BP change from baseline to day 7, and change from day 7 to day 14 will be compared
Change in fat mass and lean body mass percentage | Day 0, day 7 and day 14
  Body fat change from baseline to day 7, and change from day 7 to day 14 will be compared
Self report bias in weight, height and body fat percentage | Day 0
  Difference of measurements between self report survey and objective results
Self report of desire to lose weight and ideal weight | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil Dhurandhar, Principal Investigator — Chair of the Nutritional Sciences Department
Locations (1):
- Texas Tech University - Department of Nutritional Sciences, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bayham BE, Greenway FL, Johnson WD, Dhurandhar NV. A randomized trial to manipulate the quality instead of quantity of dietary proteins to influence the markers of satiety. J Diabetes Complications. 2014 Jul-Aug;28(4):547-52. doi: 10.1016/j.jdiacomp.2014.02.002. Epub 2014 Feb 13. PMID 24703415
- [Background] Vander Wal JS, Gupta A, Khosla P, Dhurandhar NV. Egg breakfast enhances weight loss. Int J Obes (Lond). 2008 Oct;32(10):1545-51. doi: 10.1038/ijo.2008.130. Epub 2008 Aug 5. PMID 18679412
- [Background] Vander Wal JS, Marth JM, Khosla P, Jen KL, Dhurandhar NV. Short-term effect of eggs on satiety in overweight and obese subjects. J Am Coll Nutr. 2005 Dec;24(6):510-5. doi: 10.1080/07315724.2005.10719497. PMID 16373948